CLINICAL TRIAL: NCT01309620
Title: Does Zinc Supplementation Reduce the Extent of Oxidative Stress Damage in Diabetics? A Randomised Placebo-controlled Study.
Brief Title: Zinc Supplementation in Type 2 Diabetics
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Seet Chee Seong, Raymond, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSRB A/08/045
Record Dates: First submitted 2011-03-02; First posted 2011-03-07 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: zinc, oxidative stress, vascular indices, type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — gluconic acid; Zinc

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Zinc supplement (Experimental)
  Interventions: Dietary Supplement: Zinc gluconate

INTERVENTIONS:
Dietary Supplement: Zinc gluconate — Zinc gluconate (GNC, USA), 100 mg twice daily
  Other Names: Zinc gluconate (GNC, USA); Zinc; Zinc supplementation
  Arms: Zinc supplement
Dietary Supplement: Placebo — Placebo, Twice Daily
  Arms: Placebo

SUMMARY:
Zinc supplementation reduces the extent of oxidative damage and improves vascular indices in type 2 diabetics

DETAILED DESCRIPTION:
Study participants

Forty male type 2 diabetics, recruited from the outpatient clinic at the National University Hospital, Singapore, will be randomized to receive two tablets of either 100 mg zinc gluconate (GNC, USA) or placebo (99% microcystalline cellulose, 1% magnesium stearate) per day for 3 months. Subjects aged 21 years and above who fulfilled the American Diabetes Association criteria for the diagnosis of type 2 diabetes mellitus will be included in this study. We will exclude those who: had consumed over-the counter or prescription drugs, vitamin/mineral supplements or traditional Chinese remedies, suffered acute infection less than 30-days prior to the start of the study, had been diagnosed with active neuropsychiatric disease or hematological diseases, had hemoglobin less than 10g/dL, had previous use of narcotic drugs or regular alcohol intake in excess of 14 units per week. Each participant will provide written informed consent prior to their participation in this study.

Supplementation and sampling of blood and urine

A hospital research pharmacist will be engaged to randomize, blind the assigned treatment groups and count the remaining tablets so as to assess compliance. Blood and spot urine samples will be taken following an 8-hour fast at baseline (before supplementation), days 3 and 7, months 1, 2 and 3 during supplementation and 1 month following the intake of zinc or placebo (washout). An aliquot of blood will be collected in plain or EDTA tubes for serum or plasma separation respectively.

Markers of oxidative damage

Blood samples collected into EDTA tubes will be centrifuged, indomethacin and butylated hydroxytoluene added into the plasma, and fresh urine samples placed in polypropylene tubes. The prepared samples will be stored at -80oC until analysis. Oxidative stress related biomarkers, F2-IsoPs, F4-NPs, HETEs, COPs and allantoin, will be measured by gas chromatography-mass spectrometry using methods as previously described. Briefly, mixed heavy isotopes, 8-iso-PGF2α-d4, IPF2α-VI-d4, [18O2] F4-NP (gift from Prof. Jason D. Morrow (deceased), Eiscosanoid Core Laboratory at Vanderbilt University), 5(S)-HETE-d8, 12(S)-HETE-d8, 15(S)-HETE-d8, 20-HETE-d6 and arachidonic acid-d8 and docosahexaenoic acid-d5, and 7-OH cholesterol-d7, 24-OH cholesterol-d7 and 26 (27)-OH cholesterol-d5 and 7-keto-cholesterol-d7 will be added into plasma for quantification of the oxidative stress markers. To measure the total (free and esterified) forms of F2-IsoPs, F4-NPs and HETEs products, 1 M potassium hydroxide prepared in methanol will be added to plasma (1:1) and hydrolysis performed at 37oC for 30 minutes. Thereafter, methanol, 5 M HCl and 40 mM formic acid (pH 4.6) will be sequentially added and mixed. The plasma mix will then purified using anionic exchange solid phase extraction (SPE). To measure the free forms in plasma and urine (F2-IsoPs and HETEs), 40 mM formic acid (pH 4.5) will be added to the plasma or urine sample, mixed and then purified by SPE. Urinary creatinine levels will be measured to standardize urinary F2-IsoPs and HETEs (Sigma Diagnostic kit, USA).

The purified samples will then be derivatized and analyzed using gas chromatography (Hewlett-Packard 6890, Agilent Technologies, USA) coupled to a mass selective detector (Hewlett-Packard 5973N, Agilent Technologies, USA) (GC-MS). For F2-IsoPs, F4-NPs, HETEs (a mixture of 5(S)-, 12(S)-, 15(S)- and 20-HETEs), and total arachidonate and total docosahexanoate measurements, negative chemical ionization (NCI) mode will be applied and chromatographic separations will be carried out on a fused silica capillary column coated with cross-linked 5% phenylmethylsiloxane (HP-5, Agilent Technologies, USA). To determine COPs, electron ionization mode will be applied and chromatographic separations carried out on a fused silica capillary column coated with cross-linked 5% phenylmethylsiloxane (Ultra 2 J&W, USA). Concentrations of the lipid oxidation products will be calculated by comparing the peak area of each compound with the relevant deuterated internal standard.

For allantoin and urate analysis, 25 ul plasma will be centrifuged using Nanosep filters (10 kDa) and to the filtrate, 25 ul of 4 mM 15N allantoin and 100 ul acetonitrile will be added, mixed and then dried under nitrogen gas. The dried sample will then be derivatized with 50 ml N-(butyl-dimethyl-silyl)-2,2,2-trifluoro-N-methyl-acetamide (MTBSTFA) in pyridine (1:1 v/v) at 50oC for 2 h. Allantoin will be analyzed by GC-MS. Separations will be carried out on a fused silica capillary column coated with cross-linked 5% phenylmethylsiloxane (Ultra 2, Agilent, USA). Derivatized allantoin samples (1 µl) will be injected into the GC-MS. Quantification of allantoin will be calculated by comparison with the heavy isotope.

For urate analysis, 80 ul water will be added to 20 ul plasma, mixed and then centrifuged using Nanosep filters (10 kDa). The filtrate will then be injected into an HPLC (Agilent Technologies, USA) coupled to a UV detector. Chromatographic separation will be achieved using 250 mm Zorbax SB-C8 columns under isocratic condition where 2 mM NH4H2PO4 (pH 2.95) will be used for the mobile phase. The area of the eluted uric acid peak will be measured and the concentration determined against the linear calibration curve constructed with the samples spiked with pure urate.

Clinical parameters of serum and hematological indices

Blood glucose, HbA1c and insulin, serum hsCRP, cholesterol, LDL, HDL, triglyceride and iron will be measured using the Cobas C111 analyzer (Roche Diagnostics, Switzerland). Serum zinc and copper levels will be determined at the Referral Laboratory at the Singapore General Hospital, and white and red blood counts, hemoglobin, hematocrit concentrations, platelets, neutrophils and lymphocytes, will be assessed using the Full Blood Count Analyzer (Sysmex, Japan).

Vascular indices

The technique of pulse wave analysis will be used to determine the aortic pressure and augmentation index (AIx). Pulse wave velocity recordings will be made from the radial artery using a Millar tonometer, and data will be collected and analyzed using the SphygmoCor (SphygmoCor 2000 v7.0, PWV Medical, Sydney, Australia), which allowed continuous recording of the radial artery pressure waveform. The AIx will be calculated by dividing the difference in pressure between the first and second systolic peaks of the aortic pressure waveform by the calculated aortic pulse pressure.

Measurement of plasma nitrate/nitrite will be adapted from that of Tsikas. In brief, to 200 µl of plasma heavy label 15N NO3- and 15N NO2- will be added, 800 µl acetone and 100 µl pentafluorobenzyl bromide (PFBBr) will be added, mixed and incubated at 50°C for 60 min. The acetone portion will be evaporated under nitrogen and then 500 µl of toluene will be added and mixed vigorously for 1 min. The organic extract will be obtained by centrifuging at 2000 rpm for 5 min at 4°C. Derivatized samples will be analyzed by GC-MS/NCI. Separations will be carried out on a fused silica capillary column coated with cross-linked 5% phenyl methyl siloxane. Derivatized samples (1µl) will be injected into the GC injection port using a splitless mode. Quantification of nitrate/nitrite will be calculated by comparing the peak area of each compound with the relevant heavy labelled internal standard 15N NO3- and 15N NO2-.

Statistical analyses

Statistical analysis will be performed using by GraphPad Prism version 5.0 for Macintosh (GraphPad Prism Software, CA, USA). All values will be expressed as mean SD. Paired Student's t-test will be performed between baseline and each time point during supplementation and after the wash-out period. Any significant changes detected by Student's t-test will be confirmed by ANOVA with repeated measures to assess the effects of zinc over time.

ELIGIBILITY:
Inclusion criteria:

Subjects aged 21 years and above Subjects with type 2 diabetes mellitus

Exclusion criteria:

Those who consumed over-the counter or prescription drugs, vitamin/mineral supplements or traditional Chinese remedies Those who suffered acute infection less than 30-days prior to the start of the study Those who had been diagnosed with active neuropsychiatric disease or hematological diseases Those who had hemoglobin less than 10g/dL Those who had previous use of narcotic drugs or regular alcohol intake in excess of 14 units per week.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Markers of oxidative damage | Three months
  Isoprostanes, HETEs, cholesterol oxidation products, neuroprostanes, allantoin

SECONDARY OUTCOMES:
Vascular indices | Three months
  Augmentation index and aortic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Raymond CS Seet, MBBS, Principal Investigator — National University Hospital, Singapore

REFERENCES:
- [Derived] Seet RC, Lee CY, Lim EC, Quek AM, Huang H, Huang SH, Looi WF, Long LH, Halliwell B. Oral zinc supplementation does not improve oxidative stress or vascular function in patients with type 2 diabetes with normal zinc levels. Atherosclerosis. 2011 Nov;219(1):231-9. doi: 10.1016/j.atherosclerosis.2011.07.097. Epub 2011 Jul 26. PMID 21840002